CLINICAL TRIAL: NCT05326815
Title: A Comparison of Serum and Urine N-telopeptide Marker
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-190
Record Dates: First submitted 2022-03-28; First posted 2022-04-14 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Osteoporosis; Fractures, Bone
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Osteopenia, no past medical therapy: Patients diagnosed with osteopenia on DEXA scan who have not been on any medical therapy in the past
  Interventions: Diagnostic Test: N-Telopeptide, Bone Marker

INTERVENTIONS:
Diagnostic Test: N-Telopeptide, Bone Marker — This is a prospective specimen collection cohort study to evaluate the correlation between serum and urine values of the bone marker of interest (N-Telopeptide), and their association with baseline DEXA scan measures and fracture risk within 6 months.
  Study samples will be obtained longitudinally. One collection of both serum and urine collection will be obtained. The urine will be collected as second void of day and at the same time the blood collection is drawn.

SUMMARY:
This is a prospective specimen collection cohort study to evaluate the correlation between serum and urine values of the bone marker of interest, and their association with baseline DEXA scan measures and fracture risk within 6 months.

Study samples will be obtained longitudinally. One collection of both serum and urine collection will be obtained. The urine will be collected as second void of day and at the same time the blood collection is drawn. Study will continue for a period or 1 year, with plan to enroll around 40 subjects.

DETAILED DESCRIPTION:
Osteoporosis is the most common metabolic disorder in the United States and it is estimated that approximately 19% of women and 4% of men over the age 50 years have underlying disease. This number is expected to continue to rise. A silent illness at first, once presenting with fractures, it can lead to increased morbidity, mortality, and decreased quality of life. It carries large financial and societal burdens. Direct annual medical costs are estimated to be approximately 17 to 20 billion dollars in the United States alone. Therefore, it is important to accurately identify those at high risk.

The present gold standard to diagnose osteoporosis is the Dual-energy X-ray absorptiometry (DEXA scan) with a diagnosis based on a T-score of -2.5 SD or below in those without history of fragility fracture. However, many individuals fracture despite having normal or only mildly reduced scores. There are also several barriers within the DEXA technology including accessibility, cost, accurate reference ranges for age and demographic groups that result in missing large groups of people at risk for osteoporosis. The Fracture Risk Assessment Tool (FRAX score) is one tool that identifies those at higher risk of fracture that may benefit from therapy. It was designed and released in 2008 and has been a great asset in clinical practice in stratifying risk and guiding management of osteopenic patients. However, FRAX may miss many individuals that may benefit from therapy due to its limited inclusion criteria.

Bone markers have been shown to predict fracture risk in postmenopausal women independent of bone mineral density and may help identify high risk individuals. Amino-terminal cross-linking telopeptides of type I collagen (NTX) reflects osteoclastic bone resorption. NTX can be measured in both the serum and in urine.

The accuracy of the serum NTX is unclear. It may be less sensitive than urine NTX in detecting bone density changes. The urine NTX overcomes circadian rhythm changes to bone density and is less sensitive to dietary collagen intake. At present, urine markers need to be checked as a second void of the day which may be cumbersome for patients. Serum levels drawn with other bone labs would be easier to obtain than second void urine collections. The study team involved with this research would like to evaluate the correlation between serum and urine NTX in patients with osteopenia with no prior history of osteoporotic treatment. If the urine and serum markers are equivalent methods, serum levels would be preferred to identify high risk patients at risk of disease due to ease of collection.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study
* Participants limited to subjects in the CCF
* Age between and inclusive of 18 and 85 years of age
* No gender exclusion
* Patients diagnosed with Osteopenia on DEXA scan who have not been on any medical therapy in the past
* Presence of normal vitamin D levels, kidney function, and parathyroid hormone levels (per our reference ranges)

Exclusion Criteria:

* Prior history of medical therapy for osteopenia
* Prior radiation therapy
* Prior history of bone fracture
* History of high risk medication associated with increased risk of fracture
* Presence of abnormal vitamin D levels, kidney function, and parathyroid hormone
* Pregnancy status (verbal)
* Those with medical co-morbidities that increase the risk of fracture will be excluded and these include but are not limited to: rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, diabetes mellitus, hyperparathyroidism, chronic kidney disease, pituitary disease, multiple myeloma, leukemia, lymphoma, thalassemia major, HIV/AIDS, malabsorption, Inflammatory bowel disease, chronic obstructive pulmonary disease, hypogonadism, chronic liver disease, untreated hyperthyroidism, and those with chronic immobility

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Osteopenia on DEXA scan who have not been on any medical therapy in the past Presence of normal vitamin D levels, kidney function, and parathyroid hormone levels (per our reference ranges)
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lea El Hage, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment start date- June 2022 Recruitment end date- April 2023
Pre-assignment Details: No randomization was involved with this study.
Groups:
- Osteopenia, no Past Medical Therapy: Patients diagnosed with osteopenia on DEXA scan who have not been on any medical therapy in the past
  N-Telopeptide, Bone Marker: This is a prospective specimen collection cohort study to evaluate the correlation between serum and urine values of the bone marker of interest (N-Telopeptide), and their association with baseline DEXA scan measures and fracture risk within 6 months.
  Study samples will be obtained longitudinally. One collection of both serum and urine collection will be obtained. The urine will be collected as second void of day and at the same time the blood collection is drawn.
Period: Overall Study
Arm/Group | Osteopenia, no Past Medical Therapy
Started | 54
Completed | 40
Not Completed | 14
Not completed — Withdrawal by Subject | 3
Not completed — Did not complete required labs | 6
Not completed — Screen fail- abnormal labs | 5

BASELINE CHARACTERISTICS:
Population: 14 patients who were enrolled did not complete baseline assessments
Arm/Group | Osteopenia, no Past Medical Therapy
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 36
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between NTX Measures With Each Other
Description: Correlation between NTX measures with each other
Time Frame: 1 day (single visit lab test)
Measure: Number (95% Confidence Interval); unit: r-value
Arm/Group | Osteopenia, no Past Medical Therapy
Number analyzed (Participants) | 40
r-value | 0.52 [0.25 to 0.72]
Statistical Analysis 1: Comparison: Osteopenia, no Past Medical Therapy; Test type: Other — Spearman Correlation; p < 0.001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from June 2022 until the end of study in March 2023. Patients participating on this study during a single day lab collection.
Arm/Group | Osteopenia, no Past Medical Therapy
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT05326815/Prot_SAP_000.pdf